CLINICAL TRIAL: NCT01046370
Title: A Pilot Study of Amygdala Retraining Program (ARP) Versus Control (C) in Patients With Chronic Fatigue Syndrome (CFS), Chronic Fatigue (CF) and Fibromyalgia (FM)
Brief Title: A Pilot Study of Amygdala Retraining Program in Patients With Chronic Fatigue Syndrome, Chronic Fatigue and Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ann Vincent, Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-003509
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Fatigue Syndrome; Chronic Fatigue; Fibromyalgia
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARP intervention (Experimental)
  Interventions: Behavioral: Amygdala Retraining Program
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Amygdala Retraining Program — Mind-body intervention.
  Arms: ARP intervention

SUMMARY:
The purpose of this pilot study is to gather preliminary data on the efficacy and feasibility of the Amygdala Retraining Program (ARP), a mind-body practice versus a control (C) on fatigue, quality of life and sleep in patients with Chronic Fatigue Syndrome (CFS), Chronic Fatigue (CF) and Fibromyalgia (FM).

CFS, CF and FM are incapacitating disorders characterized by profound fatigue, muscle pain, impaired memory, insomnia, and post-exertional malaise (Fukuda 1994). Current literature points to a centrally sensitized state in CFS, CF and FM (Meeus 2007). The ARP attempts to retrain this neuronal network through mind-body practices such as cognitive restructuring via neurolinguistic programming, yoga based breathing and simple mindfulness based meditation. A case series of 33 patients with CFS and ARP reported improvement in 92% of patients with two-thirds of patients reaching 80-100% of pre-illness levels of health (Gupta 2009). However ARP has never been formally studied in CFS.

We propose to gather preliminary data on the efficacy and feasibility of ARP versus C on fatigue, quality of life and sleep in 30 patients with CFS, CF and FM. All participants will undergo standard clinical treatment which consist of a 2 day self-management program in the Chronic Fatigue Clinic. Following this, participants will be randomized into the ARP or C group. The ARP group will receive an additional 2.5 hour training surrounding core concepts of the ARP program. They will then be given the ARP DVD program and booklet, to reinforce and continue the practice. They will then receive scheduled bi-monthly phone calls for 3 months from a study investigator for support. The C group will receive only standard care. However they will receive a complementary copy of the ARP program at the end of the study (6 month time point) as a gift for participation in the study.

Preliminary data on efficacy will be assessed at baseline, 1, 3 and 6 months using the following validated questionnaires: Multidimensional Fatigue Inventory (MDFI), Short form-36 (SF36) Fibromyalgia Impact Questionnaire (FIQ), Epworth Sleep Scale (ESS) and Measure Your Medical Outcome Profile (MYMOP-2). Feasibility will be assessed by evaluation of a daily practice log where patients record the total time spent daily in the practice of ARP and any specific difficulties they encountered in the practice of the program.

ELIGIBILITY:
Inclusion Criteria:

* meet CDC criteria for Chronic Fatigue Syndrome, have been diagnosed with chronic fatigue, or meet the American College of Rheumatology criteria for fibromyalgia

Exclusion Criteria:

* untreated hypo or hyper thyroidism
* untreated hypo or hyper parathyroidism
* untreated adrenal disorders
* untreated diabetes
* multiple sclerosis
* acute or chronic hepatitis
* history of cancer
* untreated depression
* chronic steroid use
* acute inflammatory rheumatological conditions
* untreated obstructive sleep apnea
* narcolepsy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
chronic fatigue syndrome, chronic fatigue and fibromyalgia symptom severity | 6 months

SECONDARY OUTCOMES:
fatigue as assessed by Multidimensional Fatigue Inventory (MDFI) and Epworth Sleep Scale (ESS) | 6 months
pain as assessed by the Fibromyalgia Impact Questionnaire (FIQ) and Measure Your Medical Outcome Profile (MYMOP-2) | 6 months
quality of life as assessed by the Short Form-36 (SF-36) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Vincent, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Toussaint LL, Whipple MO, Abboud LL, Vincent A, Wahner-Roedler DL. A mind-body technique for symptoms related to fibromyalgia and chronic fatigue. Explore (NY). 2012 Mar-Apr;8(2):92-8. doi: 10.1016/j.explore.2011.12.003. PMID 22385563